CLINICAL TRIAL: NCT05703711
Title: Combining mHealth and Nurse-delivered Care to Improve the Outcomes of People With Serious Mental Illness in West Africa
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Dror Ben-Zeev, Professor: Psychiatry & Behavioral Sciences, University of Washington
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00015549; 1R01MH127531-01A1 (NIH)
Record Dates: First submitted 2023-01-19; First posted 2023-01-30 (Actual); Last update posted 2024-07-25 (Actual); Status verified 2024-07

CONDITIONS: Psychosis; Mania; Depression
Keywords: mHealth; Psychosis; Mania; Depression
MeSH Terms: conditions — Psychotic Disorders; Mania; Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Enhanced Usual Care (No Intervention): In the Enhanced Usual Care arm, all healers are invited to participate in an interactive session reviewing ways to reduce inhumane and potentially harmful treatments in practices at their camps.
- M&M Intervention Package (Experimental): M&M is a 8-week long combination of mHealth designed to train healers to deliver basic psychosocial interventions while preserving human rights with pharmacotherapy delivered directly to their patients via visiting nurse.
  Interventions: Behavioral: mHealer

INTERVENTIONS:
Behavioral: mHealer — MHealer is a software application installed on smartphones that provides psychosocial treatment support and patient condition tracking.
  Arms: M&M Intervention Package

SUMMARY:
In West Africa, most people with serious mental illness receive care from traditional or faith healers at prayer camps. The stepped-wedge cluster randomized trial aims to evaluate the effectiveness of a dual-pronged intervention package comprised of a mobile health program designed to train healers to deliver evidence-based psychosocial interventions combined with pharmacotherapy delivered directly to the patients at their prayer camps via a visiting nurse in Ghana.

DETAILED DESCRIPTION:
The study involves deployment of an intervention in Ghanian prayer camps where traditional and faith healers provide care for people with mental illness. The intervention has two components: a visiting nurse that provides medications to patients staying at the prayer camps combined with a smartphone app called M-Healer that is used by the staff working at the camps. The app is designed to provide them with training on how to deliver some psychosocial interventions, monitor the health and well-being of their patients, and protect human rights at the camps.

The stepped-wedge cluster randomized study design involves all participant groups beginning the trial receiving enhanced usual care with random sequential crossover of groups to the experimental condition until all groups have been exposed to the full intervention. Throughout the study, participant data will be collected at baseline, mid-treatment, and post-treatment. Following study completion, the intervention will be evaluated by comparing changes in psychiatric symptoms of participants from baseline to post-treatment.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or older
* Speaks Twi or English
* Current inpatient staying at a study prayer camp
* A diagnosis of psychosis, mania, or depression

Exclusion Criteria:

* Serious physical illness or in need of urgent medical attention

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 360 (Estimated)
Dates: Start 2023-10-25 (Actual); Primary Completion 2027-05-31 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
Psychiatric symptoms | Baseline, 4 weeks, 8 weeks
  Change in psychiatric symptoms of study participants as measured by the Brief Psychiatric Rating Scale
Depressive symptoms | Baseline, 4 weeks, 8 weeks
  Change in depressive symptoms of participants as measured by the Patient Health Questionnaire-9

CONTACTS AND LOCATIONS:
Overall Officials: Dror Ben-Zeev, PhD, Principal Investigator — University of Washington
Locations (1):
- University of Ghana, Accra, Ghana

IPD SHARING:
Plan to Share IPD: Undecided
De-identified data from the study may be shared in future, yet-to-be-known, research. Data may be used to evaluate mechanism of intervention action, documentation of prevalence of psychiatric illnesses in the region, relationships between clinical or demographic variables and treatment outcomes, or use of technology in the region.